CLINICAL TRIAL: NCT05718401
Title: A Single-center Retrospective Cohort Clinical Study Was Used to Explore the Clinical Characteristics and Risk Factors of Patients With Multiple Myeloma Myocardial Amyloidosis. An Exploratory Study Was Conducted to Compare the Effects of Various Sublayer Factors on Patients' Survival. On This Basis, a Hierarchical Diagnostic Model for Patients With Multiple Myeloma Complicated With Myocardial Amyloidosis Was Established Based on the Phenoomics of NMR and Mass Spectrometry Were Evaluated Simultaneously
Brief Title: The Diagnostic Pattern and Prognosis of Multiple Myeloma Patients With Myocardial Amyloidosis Were Evaluated by NMR Based Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2022-033
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma; Amyloidosis Cardiac
MeSH Terms: conditions — Multiple Myeloma; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood or/and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Intervention group: Patients With Multiple Myeloma Myocardial Amyloidosis
  Interventions: Device: NMR
- Control group: Patients With Multiple Myeloma but without Myocardial Amyloidosis.
  Interventions: Device: NMR

INTERVENTIONS:
Device: NMR — nuclear magnetic resonance in genomics

SUMMARY:
In this clinical study, a single-center retrospective cohort study was used to explore the clinical characteristics and risk factors of patients with multiple myeloma myocardial amyloidosis. An exploratory study was conducted to compare the effects of various sublayer factors (M protein, electrocardiogram, echocardiography, CD138, chromosome abnormalities, etc.) on patients' survival. On this basis, a hierarchical diagnostic model (1-2-3-4) for patients with multiple myeloma complicated with myocardial amyloidosis was established based on the phenoomics of NMR and mass spectrometry, and the prognosis was evaluated simultaneously, in order to create an early, non-invasive, sensitive and quantitative diagnostic model for multiple myeloma complicated with myocardial amyloidosis, and lay a foundation for the early application of effective treatment.

DETAILED DESCRIPTION:
The purpose of this study was to collect clinical data of patients with multiple myeloma complicated with myocardial amyloidosis, analyze and collate the data through statistical methods, and explore the clinical characteristics of patients with MM complicated with myocardial amyloidosis, the factors that may lead to the occurrence of myocardial amyloidosis and the differences in the data of cardiac ultrasound and other biochemical tests, so as to evaluate the prognosis of patients.

To investigate the clinical features, risk factors and prognosis of patients with multiple myeloma myocardial amyloidosis. The clinical experience of diagnosis and treatment of this complication was summarized. On this basis, a standard database suitable for the northwest population was established based on NMR phenoomics, and a hierarchical diagnostic model (1-2-3-4) was explored for multiple myeloma patients with myocardial amyloidosis, and the prognosis was evaluated simultaneously. In order to establish an early, non-invasive, sensitive and quantitative diagnostic model for multiple myeloma complicated with myocardial amyloidosis, and to provide clinical basis for further research on early diagnosis, early prevention and early treatment of the disease. To provide the basis for individualized stratified prevention and treatment of patients with multiple myeloma myocardial amyloidosis, reduce the family medical burden and related side effects, improve the quality of life of patients with myeloma myocardial amyloidosis, prolong the survival period, and improve the cure rate

ELIGIBILITY:
Inclusion Criteria:

A patient with multiple myeloma complicated with myocardial amyloidosis was diagnosed in our hospital since January 1, 2018

Exclusion Criteria:

A patient without multiple myeloma complicated with myocardial amyloidosis was diagnosed in our hospital since January 1, 2018

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with multiple myeloma complicated with myocardial amyloidosis
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The long axial strain of echocardiography | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 mouths
  The long axial strain of echocardiography was in the normal range（18%-22%）

CONTACTS AND LOCATIONS:
Overall Officials: Liu huasheng, Ph.D, Study Director — First Hospital of Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi, China